CLINICAL TRIAL: NCT02916602
Title: A Randomized, Double-blind, Multicenter, Phase 3 Study to Evaluate Efficacy and Safety of HCP1401 for Stage 2 Hypertension Patients Not Controlled by HCP0605
Brief Title: A Study to Evaluate Efficacy and Safety of HCP1401 for Stage 2 Hypertension Patients Not Controlled by HCP0605
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-ALCH-301
Record Dates: First submitted 2016-09-26; First posted 2016-09-27 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; Losartan; Chlorthalidone; amlodipine-losartan drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): HCP1401
  Interventions: Drug: HCP1401
- Reference (Active Comparator): HCP0605
  Interventions: Drug: HCP0605

INTERVENTIONS:
Drug: HCP1401 — amlodipine, Losartan, Chlorthalidone FDC
  Other Names: amlodipine, Losartan, Chlorthalidone
  Arms: Treatment
Drug: HCP0605 — amlodipine, Losartan FDC
  Other Names: amlodipine, Losartan
  Arms: Reference

SUMMARY:
A phase 3 study to evaluate efficacy and safety of HCP1401

DETAILED DESCRIPTION:
A randomized, double-blind, multicenter, phase 3 study to evaluate efficacy and safety of HCP1401 for stage 2 hypertension patients not controlled by HCP0605

ELIGIBILITY:
Inclusion Criteria:

* Hypertension patient who satisfied below condition at Visit 1.

  * patient who takes antihypertensive drug

    * 140mmHg <= sitSBP <= 200mmHg
  * patient who doesn't take antihypertensive drug

    * 160mmHg <= sitSBP <= 200mmHg
    * 140mmHg <= sitSBP <= 200mmHg at Visit 2

Exclusion Criteria:

* Patient who have received 4 or more antihypertensive drug
* Patient with 20mmHg of difference in sitSBP or 10mmHg of difference in sitDBP between 3 times of BP measuring at Visit 1
* Patient with sitDBP >= 120mmHg at Visit 2
* Patient with secondary hypertension

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2015-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in sitting systolic blood pressure at week 8 | 8 weeks

SECONDARY OUTCOMES:
Change from baseline in sitting diastolic blood pressure at week 2 and week 8 | 2 weeks and 8 weeks
Change from baseline in sitting systolic blood pressure at week 2 | 2 weeks
Proportion of subjects achieving Blood Pressure control | 2 weeks and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cheulho Kim, M.D.,Ph.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hong SJ, Jeong HS, Han SH, Chang KY, Hong BK, Lee BK, Chae SC, Kim WS, Park CG, Heo JH, Lee SU, Kim YD, Kim KS, Choi JH, Kang HJ, Kim JJ, Kang SM, Choi YJ, Shin JH, Chun KJ, Shin DG, Park SH, Kwan J, Choi YJ, Jeong MH, Chae JK, Kim DW, Cho JR, Han KR, Won KH, Park SH, Lee SK, Kim SH, Jung J, Kim CH. Comparison of Fixed-dose Combinations of Amlodipine/Losartan Potassium/Chlorthalidone and Amlodipine/Losartan Potassium in Patients With Stage 2 Hypertension Inadequately Controlled With Amlodipine/Losartan Potassium: A Randomized, Double-blind, Multicenter, Phase III Study. Clin Ther. 2017 Oct;39(10):2049-2060. doi: 10.1016/j.clinthera.2017.08.013. Epub 2017 Sep 19. PMID 28939406